CLINICAL TRIAL: NCT03071055
Title: Efficacy of Biweekly Ranibizumab (0.5 mg) for Exudative Macular Degeneration Retinal Edema Refractory to Anti-VEGF Therapy Comparing Syringe Preparation Time Using Ranibizumab Vial and Pre-filled Syringe
Brief Title: Efficacy of Biweekly Ranibizumab (0.5 mg) for Exudative Macular Degeneration Retinal Edema Refractory to Anti-VEGF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southeast Clinical Research Associates, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Andrew N. Antoszyk, MD, Medical Doctor, Southeast Clinical Research Associates, LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29459
Record Dates: First submitted 2017-02-24; First posted 2017-03-06 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Exudative Age Related Macular Degeneration
Keywords: Macular Degeneration; AMD; Wet AMD; Lucentis
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ranibizumab (Active Comparator): ranibizumab 0.5mg in commercially available vial
  Interventions: Drug: Ranibizumab Injection [Lucentis]
- ranibizumab pre filled-syringe (Experimental): ranibizumab 0.5mg in soon to be available pre-filled syringe
  Interventions: Drug: Ranibizumab Injection [Lucentis]

INTERVENTIONS:
Drug: Ranibizumab Injection [Lucentis] — intravitreal injection
  Other Names: Lucentis

SUMMARY:
This is a 24 week open label study to assess the efficacy of bi-weekly ranibizumab for patients with retinal fluid due to exudative macular degeneration refractory to monthly therapy.

DETAILED DESCRIPTION:
This is a 24 week, open-label, non-randomized, phase II study evaluating intravitreal ranibizumab dosed every 14 days in subjects with exudative macular degeneration who have persistent intraretinal or subretinal fluid despite chronic monthly anti-VEGF therapy (>6 months). Subjects must have had a minimum of 5 intravitreal anti-VEGF injections administered every 4-6 weeks in the 6 months preceding enrollment.

Consented, enrolled subjects will receive multiple open-label intravitreal injections of 0.5 mg ranibizumab administered every 14 days (± 3 days). Subjects who have resolution of fluid will convert to monthly ranibizumab for the remainder of the study. If fluid recurs, subjects will return to biweekly treatment.

Patients will be assigned to receive treatment with either ranibizumab vial or PFSs so that approximately 10 patients will be treated with each delivery method option, and syringe preparation time (SPT) will be measured by an assistant who will be observing the procedure and timing with an automated stopwatch.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Exudative age related macular degeneration in study eye involving the fovea
* Best Corrected Visual Acuity (by ETDRS) letter score in study eye of < 85 and > 24 (approximate Snellen equivalent 20/20 to 20/320)
* Persistent intraretinal or subretinal fluid on SD OCT despite a minimum of 5 intravitreal anti-VEGF injections administered every 4-6 weeks in the in the 6 months preceding enrollment in the study eye
* At least 30 days from last intravitreal anti-VEGF injection in the study eye

Exclusion Criteria:

* Patient who are receiving systemic anti-VEGF or proangiogenic therapy
* Patients on chronic high doses corticosteroid therapy (> than 10 mg of oral prednisone or equivalent greater than 10 days)
* Patients on chronic immunosuppressant therapy
* Patients on drugs known to have toxic side effects on the retina e.g. hydroxychloroquine
* History of intravitreal corticosteroids in study eye within 4 months of baseline
* Uncontrolled hypertension (defined as systolic >180 mm Hg and/or diastolic > 100 mm Hg while patient is sitting)
* History of stroke or APTC event in the previous year
* Any intraocular surgery in study eye within 90 days of baseline
* Presence of vitreomacular traction in study eye
* Presence of significant epiretinal proliferation in study eye
* Evidence of active infection in either eye
* Uncontrolled glaucoma in the study eye defined as a pressure > 25 mmHg on maximal medical therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is mean change in ETDRS BCVA visual acuity | 24 weeks
  The primary outcome measure is mean change in ETDRS BCVA visual acuity at 24 weeks compared to baseline.

SECONDARY OUTCOMES:
Proportion of eyes that gain or lose >0 letters at 24 weeks | 24 weeks
  Proportion of eyes that gain or lose >0 letters at 24 weeks
Proportion of eyes that gain or lose > 5 letters at 24 weeks | 24 weeks
  Proportion of eyes that gain or lose > 5 letters at 24 weeks
Proportion of eyes that gain or lose > 10 letters at 24 weeks | 24 weeks
  Proportion of eyes that gain or lose > 10 letters at 24 weeks
Proportion of eyes that gain or lose > 15 letters at 24 weeks | 24 weeks
  Proportion of eyes that gain or lose > 15 letters at 24 weeks
To compare syringe preparation time (SPT) using ranibizumab vial and pre-filled syringe (PFS) in a real world clinical setting | 24 weeks
  To compare syringe preparation time (SPT) using ranibizumab vial and pre-filled syringe (PFS) in a real world clinical setting
• Proportion of eyes with complete resolution of subretinal fluid and/or intraretinal fluid on SD OCT (macular cube) at 24 weeks | 24 weeks
  • Proportion of eyes with complete resolution of subretinal fluid and/or intraretinal fluid on SD OCT (macular cube) at 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Charlotte Eye Ear Nose and Throat Associates, PA, Charlotte, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates, PA, Statesville, North Carolina

IPD SHARING:
Plan to Share IPD: No